CLINICAL TRIAL: NCT06434493
Title: Evaluation of Combined Modality Protons and Hepatic Transplantation for Hilar Cholangiocarcinoma (an Evaluative Commissioning in Protons Study)
Brief Title: Evaluation of Combined Modality Protons and Hepatic Transplantation for Hilar Cholangiocarcinoma
Acronym: EMPHATIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University College London Hospitals (Other); University College, London (Other); Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFTSp218 (02)
Record Dates: First submitted 2024-04-25; First posted 2024-05-30 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-05

CONDITIONS: Cholangiocarcinoma
Keywords: proton beam therapy; protons; evaluative commissioning; liver transplant
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Proton Therapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proton Beam Therapy (Experimental): All patients to be offered neoadjuvant proton beam therapy to a dose of 45 Gray (Gy) in 15 fractions over 3 weeks, with a tumour boost to 67.5 Gray (Gy), and alongside concurrent oral capecitabine 625mg/m2 twice daily on radiation days.
  Interventions: Radiation: Proton Beam Therapy; Drug: Concurrent oral capecitabine chemotherapy; Drug: Cisplatin & Gemcitabine intravenous chemotherapy; Procedure: Orthotropic Liver Transplant

INTERVENTIONS:
Radiation: Proton Beam Therapy — All patients to be offered neoadjuvant proton beam therapy to a dose of 45 Gray (Gy) in 15 fractions over 3 weeks, with a tumour boost to 67.5 Gray (Gy)
Drug: Concurrent oral capecitabine chemotherapy — All patients to be offered concurrent oral capecitabine 625mg/m2 twice daily on radiation days
Drug: Cisplatin & Gemcitabine intravenous chemotherapy — Following chemoradiotherapy (PBT + capecitabine), and whilst on the liver transplant waiting list, patients will be offered up to 6 cycles of standard chemotherapy with cisplatin and gemcitabine.
Procedure: Orthotropic Liver Transplant — If still eligible after neoadjuvant treatment (PBT + capecitabine), patients will be added to the liver transplant waiting list.

SUMMARY:
Proton Beam Therapy (PBT) is an advanced radiotherapy technique. There are two National Health Service (NHS) PBT treatment centres in the United Kingdom (UK), in Manchester and London. The NHS is committed to ensuring the best use of this limited resource by investigating which patients will benefit from PBT.

Evaluative Commissioning in Protons (ECIP) is a programme of studies exploring the role of PBT in different types of cancer. The studies are funded by NHS England. ECIP studies are not randomised studies, which means that all eligible patients will be offered PBT. Any eligible patient in the UK can be referred, and accommodation is available for patients who don't live close to a PBT centre.

The main benefit of PBT, compared with standard photon radiotherapy, is the predicted reduction in radiation dose to surrounding healthy tissues. With photon radiotherapy, some radiation passes beyond the target area, affecting healthy tissues and causing side-effects. With PBT, the radiation dose stops within the target area, causing less damage to surrounding tissues, and limiting side effects.

EMPHATIC is a study within the ECIP programme. In EMPHATIC, the investigators are looking to see whether a combination of treatments, including PBT, chemotherapy and a liver transplant, can be used to treat patients with cholangiocarcinoma (bile duct cancer).

EMPHATIC offers patients whose cancer can't be removed with surgery (unresectable) a potentially curative treatment option. There is evidence that liver transplant is a curative treatment option in patients with cholangiocarcinoma. There is a risk that the cancer may grow or spread whilst waiting for a transplant, potentially making patients ineligible. PBT and chemotherapy is thought to be the best way to control the cancer, until a liver transplant can be performed. EMPHATIC will look at how a combination of PBT and chemotherapy, followed by a liver transplant, can be used to curatively treat patients with unresectable cholangiocarcinomas.

DETAILED DESCRIPTION:
Liver and bile duct resection with lymphadenectomy is the standard of care for patients with hilar cholangiocarcinoma. Unfortunately, resection is only possible in a minority of patients for many reasons including, the extent of cancer or the presence of background primary sclerosing cholangitis (PSC). For patients with a background of PSC, liver transplantation is a potential treatment, and it was recently approved as an indication for a commissioned pilot service evaluation of liver transplantation in the UK.

Until recently, the use of liver transplantation for hilar cholangiocarcinoma was confined to a few centres in the United States. The initial publications from the Mayo Clinic and Nebraska, as well as more recent experience from other centres, support strict selection protocols to identify patients likely to benefit from liver transplantation. In 2000, the initial experience at the Mayo Clinic in which 19 patients enrolled in a pre-transplant neoadjuvant therapy protocol was published. 11 patients underwent subsequent liver transplantation. Of the 8 with long term follow up (median 44 months), only one patient developed cancer recurrence. Similarly, the long-term experience of patients in Nebraska, where 11 patients underwent liver transplantation after neoadjuvant chemoradiotherapy was published in 2002. 5 of the 11 patients were alive and disease free at a median follow up of 7.5 years .

Most recent experience is based on adopting the Mayo protocol. In general, the inclusion criteria define patients with early cancers, with a dominant stricture or tumour less than 3cm. Intra and extrahepatic disease including any site of nodal metastases precluded selection. Controversially, histology or cytology was not considered essential for diagnosis of cholangiocarcinoma by most centres. Elevated Ca 19.9 of >100, Fluorescence In Situ Hybridization (FISH) polysomy 9p21 or tumour mass in the presence of a dominant stricture were considered sufficient for enrolment. Prior (attempts at) trans-peritoneal biopsy was another exclusion criterion based on concerns of increased risk of tumour dissemination. Neoadjuvant therapy involved external beam radiation therapy (EBRT) with concurrent chemotherapy (chemo sensitisation), followed by brachytherapy whenever possible. Patients were then re-staged and remain on systemic chemotherapy until the time of transplant.

A recent review looked at all studies from 2000 until 2019. 20 studies with 428 patients were eligible for analysis. The pooled 1, 3-, and 5-year overall survival rates following liver transplantation without neoadjuvant therapy (n=156) were 71.2%. In patients who had neoadjuvant therapy prior to transplantation (n=272), the survival improved to 82.8% at 1,3 and 5 years respectively.

The cancer recurrence rate was 51.7% in patients who did not receive neoadjuvant therapy compared to 24.1% for patients who had. Only 4 of the 20 studies reported pre-transplant histological confirmation of adenocarcinoma or malignant/suspicious cells on cytology. 98% of liver explants from studies not using neoadjuvant therapy confirmed malignancy, compared to 50.5% in those who had received neoadjuvant therapy. Patients in whom malignancy was not found are presumed to have had complete pathological response to neoadjuvant therapy (approximately 50% following neoadjuvant therapy). Patients with background PSC had better outcomes compared to patients with de novo cancers.

Study Design & development of an evaluative commissioning study within ECIP:

It is not possible to design EMPHATIC, a study for patients with unresectable cholangiocarcinoma, as a randomised controlled trial (RCT), because there is no ethically acceptable control arm. In an RCT, patients in a theoretical control arm would be offered either no transplant, or no neoadjuvant therapy prior to the transplant. Based on the published literature summarised above, the adverse anticipated outcomes of patients in such a control arm would not be considered justified.

Neoadjuvant therapy is required to control the tumour prior to transplant. In the Mayo protocol described above, patients received external beam (chemo)radiotherapy followed by brachytherapy, and thereafter received chemotherapy until the time of transplant. Unfortunately, in the UK, brachytherapy services were not seen as a viable option, and hence the Mayo protocol is not feasible.

There is good scientific rationale that proton beam radiotherapy (PBT) offers the optimal technique for delivering neoadjuvant therapy as it is non-invasive, and spares as much functional liver as possible, compared with alternatives such as photon-EBRT techniques or invasive techniques (e.g. brachytherapy). Compared with photon-EBRT techniques, PBT delivers highly conformal radiotherapy, with a significantly reduced integral body dose, and no exit beam. It is expected to be associated with an improved toxicity profile.

ELIGIBILITY:
Inclusion Criteria:

General criteria

* Age 17 years and over
* Performance status 0 or 1 (Eastern Cooperative Oncology Group)
* Suitable for liver transplantation as determined by Multi Disciplinary Team (MDT)
* Able to tolerate neoadjuvant therapy.
* A history of primary sclerosing cholangitis (PSC) will be a necessary eligibility criterion at the start of the study. Part-way through recruitment to the study, the eligibility criteria may be broadened, allowing patients with sporadic / non-PSC unresectable cholangiocarcinoma to also be considered. The decision to do this will be taken by the Study Management Group, who will be monitor results closely, following an interim analysis after the first 10 patients. Suitability for Orthotropic Liver Transplant will continue to be confirmed in the regional Hepato Biliary cancer MDT.

Specific criteria

* Presence of a dominant hilar stricture or mass <3cm on cross-sectional imaging
* Histologically proven cholangiocarcinoma by brush cytology or biopsy via Endoscopic Retrograde Cholangiopancreatography (ERCP) or Percutaneous Transhepatic Cholangiography (PTC)
* No metastatic disease, including to regional lymph nodes.

Exclusion Criteria:

General criteria

* Inability to consent
* Poor performance status
* Failed fitness assessment
* Extrahepatic disease at any stage of presentation, assessment and treatment
* Prior biliary resection or hilar dissection for attempted resection within the past 12 months
* Prior malignancy in the last 5 years (excluding early breast, prostate, cervix and non melanoma skin cancers)

Specific criteria

* Estimated Glomerular Filtration Rate (eGFR) <30
* Prior radiation to the upper abdomen
* Uncontrolled infection
* Duodenal invasion

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Common Toxicity Criteria for recording Adverse Events (CTCAE) Grade 3 and above toxicity | Up to 90 days post neoadjuvant chemo-radiation.
  Incidence of Grade ≥ 3 toxicity using CTCAE (grades 0-5) up to 90 days following completion of neoadjuvant (chemo)-PBT and liver transplant. Higher score indicates worse outcome.
Proportion of patients who undergo a successful liver transplant | 90 days post transplant.
  The proportion of patients who, following neoadjuvant (chemo)-PBT, undergo a successful liver transplant (measured at 90 days post-transplant).

SECONDARY OUTCOMES:
Number of patients completing planned radiotherapy | Up to 1 year
  Number of patients completing planned radiotherapy
Incidence of severe treatment related side effects | Up to 2 years
  Rate of Common Toxicity Criteria for recording Adverse Events (CTCAE) Grade 3 and above toxicity (Grades 0-5). Higher score may mean a worse outcome.
1 year post completion of neoadjuvant therapy cancer-related mortality | At 1 year
  Calculated from date of last PBT treatment and defined as time to death or censoring at 1 year.
1 year post transplant overall survival | At 1 year
  Calculated from date of liver transplant and defined as time to death or censoring at 1 year.
1 year post transplant graft survival | At 1 year
  Calculated from date of transplant and defined as time to death or censoring at 1 year.
1 year post listing patient survival | At 1 year
  Calculated from the date the patient was added to the transplant waiting list and defined as time to death or censoring at 1 year.
Disease free survival from transplant | At 1 year
  Calculated as time to cancer recurrence or death whichever is earliest, from date of transplant, with censoring at 1 year.
Recurrent cancer within 6 months of transplant | Up to 6 months following transplant
  Described as local, regional or metastatic disease
Cancer control at time of transplant | Up to 2 years
  Reported as time to loss of cancer control with censoring at time of transplant
Cancer control at time of removal from transplant list | Up to 2 years
  Reported as time to loss of cancer control with censoring at date of removal from transplant waiting list
Transplant complication rates | Within 3 months of surgery
  Surgical complication rates according to Clavien Dindo scale, measured from grades 1-5, higher grade may mean worse outcome.
Patient pathway | Up to 2 years
  Review of patient pathway deliverability defined as time interval from patient referral to the start of chemo-PBT treatment
Time to completion of neoadjuvant chemo-PBT treatment to liver transplant | Up to 2 years
  Measured in days from last day of PBT to date of transplant
Time spent on transplant waiting list | Up to 2 years
  Measured in weeks from transplant listing date to liver transplant date
Referral rates | At 6 months, 12 months, 18 months and 24 months following the opening of the study
  Review annual referral rates to the study
Recruitment rates | At 6 months, 12 months, 18 months and 24 months following the opening of the study
  Number of patients participating in the study

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hawkins, Principal Investigator — University College, London; Douglas Thorburn, Principal Investigator — The Royal Free NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Vreede I, Steers JL, Burch PA, Rosen CB, Gunderson LL, Haddock MG, Burgart L, Gores GJ. Prolonged disease-free survival after orthotopic liver transplantation plus adjuvant chemoirradiation for cholangiocarcinoma. Liver Transpl. 2000 May;6(3):309-16. doi: 10.1053/lv.2000.6143. PMID 10827231
- [Background] Sudan D, DeRoover A, Chinnakotla S, Fox I, Shaw B Jr, McCashland T, Sorrell M, Tempero M, Langnas A. Radiochemotherapy and transplantation allow long-term survival for nonresectable hilar cholangiocarcinoma. Am J Transplant. 2002 Sep;2(8):774-9. doi: 10.1034/j.1600-6143.2002.20812.x. PMID 12243499
- [Background] Cambridge WA, Fairfield C, Powell JJ, Harrison EM, Soreide K, Wigmore SJ, Guest RV. Meta-analysis and Meta-regression of Survival After Liver Transplantation for Unresectable Perihilar Cholangiocarcinoma. Ann Surg. 2021 Feb 1;273(2):240-250. doi: 10.1097/SLA.0000000000003801. PMID 32097164